CLINICAL TRIAL: NCT05478967
Title: The Effect of Adjunctive Intravitreal Aflibercept for Preventing Postvitrectomy Hemorrhage in Proliferative Diabetic Retinopathy
Brief Title: The Effect of IVA for Preventing Postvitrectomy Hemorrhage in PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai 10th People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Nanjing Medical University (Other); Xiamen University (Other)
Responsible Party: Principal Investigator, Jinfeng Qu, Clinical Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IVAPDR
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; vitrectomy; Aflibercept; intravitreal injection; postvitrectomy hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVA group (Experimental): Received an IVA (0.5 mg/0.05 ml) injection before surgery (1 to 5 days before surgery)
  Interventions: Procedure: IVA injection before vitrectomy
- control group (No Intervention): Did not receive IVA injection before vitrectomy

INTERVENTIONS:
Procedure: IVA injection before vitrectomy — Patients in IVA group received an IVA (0.5 mg/0.05 ml) injection before surgery (1 to 5 days before surgery)
  Arms: IVA group

SUMMARY:
Aflibercept, a recombinant fusion antibody that binds to all subtypes of VEGF and PlGF, has been shown to induce effective regression of retinal neovascularization secondary to PDR but there had been lack of a well-structured prospective study about adjunctive use of intravitreal injection of Aflibercept (IVA) to reduce postoperative VH in PPV for PDR. In this study, we aim to assess the effect of preoperative IVA on the incidence of postoperative VH after PPV for PDR.

DETAILED DESCRIPTION:
The enrolled eyes were randomly assigned according to the Central Randomization System with a ratio of 1∶1 to IVA group and control group. Patients in IVA group received an IVA (0.5 mg/0.05 ml) injection before surgery (1 to 5 days before surgery); patients in control group did not receive IVA injection before vitrectomy. The preoperative IVA injection was performed following a standard protocol. All patients underwent 25-gauge transconjunctival sutureless vitrectomy using the 25-gauge trocar and cannula system under local or anesthesia. Procedures such as fibrovascular membrane dissection, endodiathermy, or endolaser photocoagulation were performed with 25-gauge instruments as required. Intraoperative bleeding was controlled by either endodiathermy or increasing the irrigation pressure. Patients were examined 1 week, 1 month, 2 months, and 3 months after surgery if there were no postoperative events. If postoperative complications, including VH, occurred, patients were instructed to visit the clinic regardless of the visit schedule. At each visit, any events involving the study eye between the visit schedules were recorded accordingly. At each postoperative visit, slit-lamp biomicroscope, indirect ophthalmoscopy, and fundus photographs were performed. The primary outcome of this study was incidence of VH after vitrectomy.

Postoperative VH was defined as a new episode of VH of grade 1 or above occurring later than 3 days after primary surgery and was evaluated according to the Diabetic Retinopathy Vitrectomy Study grading system. Incidence of VH at week 1, month 1, month 2 and month 3 were recorded. In the case of gas-injected eye, complications were assessed in the region without the gas bubble.

Preoperative, intraoperative, and postoperative data were collected for each patient. Preoperative data included age; sex; duration and status of diabetes mellitus (HbA1C); other systemic diseases such as hypertension and renal function (serum creatinine); and ophthalmic parameters including best-corrected visual acuity (BCVA), intraocular pressure (IOP), lens status, previous pan-retinal photocoagulation (PRP), and indication for surgery. Intraoperative data included phacoemulsification and intraocular lens (IOL) procedures, SF6 or air tamponade, and the presence of fibrovascular proliferation and tractional retinal detachment. Postoperative data included BCVA at each visit and number of episodes of complications.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* age between 35 and 65
* PDR who underwent primary pars plana vitrectomy for VH.

Exclusion Criteria:

* eyes with retinal tear
* eyes with iris or anterior angle neovascularization
* eyes with intraoperative use of silicone oil
* eyes with choroidal or retinal disease other than PDR or any inflammation condition
* eyes underwent any previous vitrectomy or scleral buckle surgery
* eyes received intraocular TA injection within 90 days before screening
* eyes received intraocular anti VEGF treatment within 60 days before screening or contralateral eyes received intraocular anti VEGF treatment during follow-up
* patients who had taken aspirin orally within 7 days before screening
* patient has coagulation mechanism disorder or other medicine for anticoagulant treatment
* cerebrovascular accident and / or myocardial infarction occurred within 180 days before screening
* patients with uncontrolled blood pressure (sitting position > 160 / 100 mmHg)
* patients with liver or kidney dysfunction or any severe systemic disease.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of VH | one month after vitrectomy
  Postoperative VH was defined as a new episode of VH of grade 1 or above occurring later than 3 days after primary surgery and was evaluated according to the Diabetic Retinopathy Vitrectomy Study grading system.

SECONDARY OUTCOMES:
Changes of BCVA | 1 week, 1 month, 2 months and 3 months after vitrectomy
  Changes of BCVA （LogMAR）from baseline at 1 week, 1 month, 2 months and 3 months after vitrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No